CLINICAL TRIAL: NCT02361593
Title: Transparent Cap-assisted Endoscopic Sclerotherapy(Lauromacrogol Injection) in Esophageal Varices: a Randomized Controlled Trial
Brief Title: Transparent Cap-assisted Endoscopic Sclerotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAP-VARICE
Record Dates: First submitted 2015-01-24; First posted 2015-02-12 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Esophageal Varices
Keywords: endoscopic sclerotherapy, esophageal varices, transparent cap
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cap group (Experimental): Patients will receive endoscopic sclerotherapy(lauromacrogol injection) for esophageal varices with assistance of a transparent cap in front of gastroscopy.
  Interventions: Procedure: assistance of a transparent cap
- Control group (Active Comparator): Patients will receive routine endoscopic sclerotherapy(lauromacrogol injection) for esophageal varices(no transparent cap involved).
  Interventions: Procedure: without a transparent cap

INTERVENTIONS:
Procedure: assistance of a transparent cap — Patients will receive endoscopic injection of lauromacrogol with assistance of a transparent cap.
  Arms: Cap group
Procedure: without a transparent cap — Patients will receive routine endoscopic injection of lauromacrogol without use of transparent cap.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate efficacy and safety of transparent cap-assisted endoscopic sclerotherapyI(lauromacrogol injection) in management of esophageal varices.

DETAILED DESCRIPTION:
Endoscopic procedures now play a great role in management of esophagogastric varices. Endoscopic variceal ligation(EVL) was recommended as first line therapy for primary and secondary prophylaxis in patients with esophageal varices. Previous studies have showed a superiority of EVL over endoscopic injection of sclerotherapy(EIS), mainly because of lower occurrence rate of complications. Procedure related complications were related to total amount of lauromacrogol, number of treatment and expertise of the endoscopists. Transparent cap has already been reported to assist in other endoscopic procedures, such as biopsy of Barret esophagus or endoscopic submucosal dissection. Accuracy and vision were improved with the help of transparent cap in the front of endoscopy. We have tried transparent cap-assisted sclerotherapy in some patients with in our hospital. Now a randomized controlled trial was conducted to evaluate efficacy and safety of transparent cap-assisted endoscopic sclerotherapy in management of esophageal varices.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented to our hospital with esophageal varices diagnosed by gastroscopy, with or without gastric varices.
* The age of the patients range from 18 to 80 years old.

Exclusion Criteria:

* Patients who have contraindications for lauromacrogol therapy or transparent cap.
* Patients who have no previous upper gastrointestinal bleeding history.
* Patients who have fecal disease that could greatly impact survival, such as uremia, advanced cancer or respiratory failure, et al.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
rebleeding rate | From date of randomization until the date of first rebleeding episode, assessed up to 1 month
  Rebleeding was defined as melena or hematemasis

SECONDARY OUTCOMES:
incidence rate of complications | From date of randomization until 1 month after randomization
  Participants will be followed for up to 1 month starting from the date of enrollment.Complications associated with endoscopic treatments include transient fever, transient dysphagia, transient arrhythmias, ulceration, perforation, stricture, rebleeding, aspiration pneumonia, sepsis, peritonitis and chest pain.
mortality rate | From date of randomization until the date of death, assessed up to 1 month
  Patients will be followed up for 1 month and all-cause death will be recorded.
time consumption of the procedure | From the beginning of the endoscopic injection until the end of the procedure.
occurrence rate of bleeding during the procedure | From the beginning of the endoscopic injection, until the end of the procedure.
  Bleeding was defined as visible errhysis seen from gastroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao CHEN, M.D., Study Director — Zhongshan Hospital, Shanghai
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China